CLINICAL TRIAL: NCT07266441
Title: A Phase 2, Open-label Study of JNJ-79635322 in Participants With Relapsed or Refractory Multiple Myeloma (RRMM) Who Have Received at Least 3 Prior Lines of Therapy Including a PI, an IMiD, and an Anti-CD38 Antibody
Brief Title: A Study of JNJ-79635322 in Participants With Relapsed or Refractory Multiple Myeloma
Acronym: TRIlogy-3
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 79635322MMY2001; 79635322MMY2001 (Other: Janssen Research & Development, LLC); 2025-521976-80-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- JNJ-79635322 (Experimental): Participants will receive JNJ-79635322 as an injection under the skin.
  Interventions: Drug: JNJ-79635322

INTERVENTIONS:
Drug: JNJ-79635322 — JNJ-79635322 will be administered as an injection under the skin.

SUMMARY:
The purpose of this study is to evaluate how well JNJ-79635322 works (efficacy) in participants with Relapsed or Refractory Multiple Myeloma (RRMM; a cancer that forms in a type of white blood cells called a plasma cell. Cancer is called relapsed if it comes back after treatment and is called 'refractory' if does not respond to treatment) who have received at least 3 prior lines of therapy.

ELIGIBILITY:
Inclusion:

* Documented diagnosis of multiple myeloma (MM) as defined by the criteria below:

  1. MM diagnosis according to the international myeloma working group (IMWG) diagnostic criteria
  2. Measurable disease at screening as assessed by central laboratory
* Received at least 3 prior lines of antimyeloma therapy including a proteasome inhibitor (PI), an immunomodulatory drug (IMiD), and an anti-cluster of differentiation (CD) 38 monoclonal antibody (mAb)
* Documented evidence of progressive disease(PD) or failure to achieve a response to the last line of therapy based on investigator's determination of response by the IMWG criteria
* Have discontinued concurrent use of any other anticancer treatment (including nonpalliative radiotherapy) or investigational agent
* Have an eastern cooperative oncology group (ECOG) performance status (PS) of 0 to 2 at screening and immediately before the start of study treatment administration

Exclusion:

* Suspected or known allergies, hypersensitivity, or intolerance to excipients of JNJ-79635322
* Had major surgery within 2 weeks before first dose or has planned major surgery during study treatment phase
* Known active or prior central nervous system (CNS) involvement or exhibits clinical signs of meningeal involvement of MM
* Participant has leptomeningeal disease
* Participant has a prior or concurrent second malignancy the natural history or treatment of which could likely interfere with any study endpoints of safety or the efficacy of the study treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 157 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2027-06-14 (Estimated); Study Completion 2028-12-12 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Up to 2 years and 9 months

SECONDARY OUTCOMES:
Very Good Partial Response (VGPR) or Better Rate | Up to 2 years and 9 months
Complete Response (CR) or Better Rate | Up to 2 years and 9 months
Duration of Response (DoR) | Up to 2 years and 9 months
Progression-Free Survival (PFS) | Up to 2 years and 9 months
Overall Survival (OS) | Up to 2 years and 9 months
Time To Next Line of Therapy (TTNT) | Up to 2 years and 9 months
Number of Participants With Treatment-Emergent Adverse Event (TEAE) by Severity | Up to 2 years and 9 months
Change from Baseline in Symptoms, Functioning, and Health-related Quality of Life (HRQoL) as Assessed by Multiple Myeloma Symptom and Impact Questionnaire (MySIm-Q) Scale Score | From Baseline up to 2 years and 9 months
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by European Organization for Research and Treatment of Cancer Quality of life Questionnaire Core 30 (EORTC-QLQ-C30) Scale Score | From Baseline up to 2 years and 9 months
Change from Baseline in Symptoms, Functioning, and HRQoL as Assessed by European Quality of Life 5-Dimensions 5-Level Version (EQ-5D-5L) Scale Score | From Baseline up to 2 years and 9 months
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by MySIm-Q | Up to 2 years and 9 months
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by EORTC-QLQ-C30 | Up to 2 years and 9 months
Time to Worsening in Symptoms, Functioning, and HRQoL as Assessed by EQ-5D-5L | Up to 2 years and 9 months
Percentage of Participants With Meaningful Improvement in Symptoms, Functioning, and HRQoL as Assessed by MySIm-Q | Up to 2 years and 9 months
Percentage of Participants With Meaningful Improvement in Symptoms, Functioning, and HRQoL as Assessed by EORTC-QLQ-C30 | Up to 2 years and 9 months
Percentage of Participants With Meaningful Improvement in Symptoms, Functioning, and HRQoL as Assessed by EQ-5D-5L | Up to 2 years and 9 months
Serum Concentrations for JNJ-79635322 | Up to 2 years and 9 months
Number of Participants With Anti JNJ-79635322 Antibodies | Up to 2 years and 9 months
Number of Participants With JNJ-79635322 Neutralizing Antibodies (NAb) | Up to 2 years and 9 months

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of Johnson & Johnson Innovative Medicine is available at innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu
URL: https://innovativemedicine.jnj.com/our-innovation/clinical-trials/transparency